CLINICAL TRIAL: NCT00072319
Title: Pilot Study of Epirubicin and Cyclophosphamide Followed by Paclitaxel at 10-11 Days Interval for Women With Early Breast Carcinoma
Brief Title: Neoadjuvant or Adjuvant Epirubicin, Cyclophosphamide, and Paclitaxel in Treating Women With Stage I, Stage II, or Stage III Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Pharmacia (Industry); Amgen (Industry)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: 03-092; P30CA008748 (NIH); MSKCC-03092
Record Dates: First submitted 2003-11-04; First posted 2003-11-06 (Estimated); Last update posted 2013-03-04 (Estimated); Status verified 2013-03

CONDITIONS: Breast Cancer
Keywords: stage I breast cancer; stage II breast cancer; stage IIIA breast cancer; stage IIIB breast cancer; stage IIIC breast cancer; inflammatory breast cancer
MeSH Terms: conditions — Breast Neoplasms; Inflammatory Breast Neoplasms | interventions — Filgrastim; Cyclophosphamide; Epirubicin; Paclitaxel; Chemotherapy, Adjuvant; Neoadjuvant Therapy

INTERVENTIONS:
Biological: filgrastim
Drug: cyclophosphamide
Drug: epirubicin hydrochloride
Drug: paclitaxel
Procedure: adjuvant therapy
Procedure: neoadjuvant therapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as epirubicin, cyclophosphamide, and paclitaxel, use different ways to stop tumor cells from dividing so they stop growing or die. Giving chemotherapy drugs before surgery may shrink the tumor so that it can be removed during surgery. Giving chemotherapy drugs after surgery may kill any remaining tumor cells.

PURPOSE: Pilot trial to study the effectiveness of neoadjuvant or adjuvant epirubicin, cyclophosphamide, and paclitaxel in treating women who have stage I, stage II, or stage III breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the feasibility and safety of neoadjuvant or adjuvant epirubicin, cyclophosphamide, and paclitaxel, in terms of the absence of any grade 3 or higher toxicity (aside from alopecia), in women with high-risk stage I-III breast cancer.

OUTLINE: This is a pilot study.

* Neoadjuvant or adjuvant EC therapy: Patients receive epirubicin IV over 3-5 minutes and cyclophosphamide IV (EC) on day 1 and filgrastim (G-CSF) subcutaneously on days 2-9 or 10. Treatment repeats every 10-11 days for 4 courses in the absence of disease progression or unacceptable toxicity.
* Neoadjuvant or adjuvant paclitaxel therapy: After the completion of EC therapy, patients receive paclitaxel IV over 3 hours on day 1. Patients also receive G-CSF as in EC therapy. Treatment repeats every 10-11 days for 4 courses in the absence of disease progression or unacceptable toxicity.

Patients who have not had prior surgery undergo definitive surgery after the completion of chemotherapy. Patients also may receive adjuvant radiotherapy and/or hormonal therapy at the discretion of the treating physician.

Patients are followed every 4 months for 3 years and then every 6 months for 2 years.

PROJECTED ACCRUAL: A total of 11-38 patients will be accrued for this study within 1 year.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed adenocarcinoma of the breast

  * Stage I, II, or III
  * Inflammatory breast cancer allowed
* Hormone receptor status:

  * Not specified

PATIENT CHARACTERISTICS:

Age

* 18 and over

Sex

* Female

Menopausal status

* Not specified

Performance status

* ECOG 0-1

Life expectancy

* Not specified

Hematopoietic

* Absolute neutrophil count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3

Hepatic

* Bilirubin normal
* SGOT/SGPT no greater than 2.5 times upper limit of normal (ULN) AND alkaline phosphatase no greater than ULN OR
* SGOT/SGPT no greater than ULN AND alkaline phosphatase no greater than 4 times ULN

Renal

* Not specified

Cardiovascular

* LVEF at least lower limit of normal by MUGA or echocardiogram
* No unstable angina
* No congestive heart failure
* No arrhythmia requiring medical therapy
* No myocardial infarction within the past year

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No prior allergy/hypersensitivity to any of the study drugs or other drugs formulated with Cremophor EL
* No psychiatric illness that would preclude understanding of the nature of the study or study compliance
* No active unresolved infection
* No peripheral neuropathy greater than grade 1
* No other nonmammary malignancy within the past 5 years except adequately treated nonmelanoma skin cancer or carcinoma in situ of the cervix
* No concurrent medical condition that would preclude study participation in the judgment of the investigator

PRIOR CONCURRENT THERAPY:

Biologic therapy

* More than 12 months since prior immunotherapy for prior breast cancer
* No prior or concurrent biologic therapy or immunotherapy for this breast cancer

Chemotherapy

* More than 12 months since prior chemotherapy for prior breast cancer
* No prior anthracycline (i.e., doxorubicin or epirubicin) and taxane therapy
* No prior or other concurrent chemotherapy for this breast cancer

Endocrine therapy

* No concurrent hormonal therapy for chemoprevention

  * Prior hormonal therapy for chemoprevention allowed
* No concurrent sex hormonal therapy (e.g., birth control pills or ovarian hormonal replacement therapy)

Radiotherapy

* No prior radiotherapy
* No other concurrent radiotherapy for this breast cancer

Surgery

* Not specified

Other

* No concurrent digitalis, beta-blockers, or calcium channel blockers for congestive heart failure

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2003-08; Primary Completion 2006-11 (Actual); Study Completion 2006-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Monica N. Fornier, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States